CLINICAL TRIAL: NCT03632928
Title: Day to Day Variation of Pressure Pain Threshold and Muscle Hardness in Migraine Patients
Brief Title: Day to Day Variation of Pressure Pain Threshold and Muscle Hardness
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Jeppe Hvedstrup Mann, MD., Clinical assistant, PhD Student, Danish Headache Center
Other Study IDs: 002
Record Dates: First submitted 2018-06-05; First posted 2018-08-16 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Migraine Disorders; Tenderness, Muscle; Headache Disorders
Keywords: Ultrasound elastography; Pressure pain threshold; variation
MeSH Terms: conditions — Migraine Disorders; Myalgia; Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Migraine patients: Migraine patients, who do not have any other diseases except from tension type headache.
  No intervention, but daily measurements of muscle hardness (Ultrasound Elastography) and tenderness (Pressure pain threshold)
  Interventions: Other: Ultrasound Elastography; Other: Pressure Pain threshold

INTERVENTIONS:
Other: Ultrasound Elastography — Measuring muscle hardness at the trapezius and neck bilateral
Other: Pressure Pain threshold — Measuring Pressure pain threshold at the trapezius and neck bilateral

SUMMARY:
The aim is to establish how headache and migraine can affect muscle hardness and tenderness in migraine patients

DETAILED DESCRIPTION:
Migraine is a very common disorder, and many migraine patients have symptoms from their neck and muscles. 50% of migraine patients have a sensation of stiff neck in relation to migraine attacks. Furthermore it is well established, that migraine patients have tender muscles during migraine attack, which can be measured with pressure pain threshold.

In this study the investigators aim to establish the variation in ultrasound elastography and pressure pain threshold in migraine patients over time. And establish the significance of headache, migraine and prodromes on these measurements.

The study includes daily measurements of muscle hardness and muscle tenderness. The patients are asked to fulfill a headache diary and a short questionnaire asking about current headache, physical activity, stress and current infectious diseases. Sleep and physical activity is also measured objectively using a fitbit Charge2. Furthermore the patients are asked about symptoms which often are associated with migraine (prodromes).

ELIGIBILITY:
Inclusion Criteria:

* Migraine Patient fulfilling international classification of headache disorders (ICHD 3) criteria

Exclusion Criteria:

* regular medication use other than medication for migraine or headache
* Other Pain disorders
* Musculoskeletal disorders affecting neck or upper body

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Migraine patients fulfilling the ICHD 3 Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Effect of migraine on muscle tenderness | Daily measurements for about 30-60 days in a row
  Muscle tenderness will be measured every day with pressure pain threshold. Migraine and headache is noted in a headache diary.
  Is the next measurement of muscle tenderness after migraine attack higher than those with out temporal proximity to headache. (paired T-test)
Effect of migraine on muscle hardness | Daily measurements for about 30-60 days in a row
  Muscle hardness will be measured every day with Ultrasound elastography. Migraine and headache is noted in a headache diary.
  Is the next measurement of muscle tenderness after migraine attack higher than those with out temporal proximity to headache. (paired T-test)
Regression analysis of muscle hardness | Daily measurements for about 30-60 days in a row
  Muscle hardness as the dependent variable and the following as the independent variables: Current migraine, Days until next migraine attack, days since last migraine attack, Sleep quality, physical activity, Stiff Neck (subjective feeling).
  The result shows how much of the variability in muscle hardness that can be explained by the independent variables.
Regression analysis of muscle tenderness | Daily measurements for about 30-60 days in a row
  Muscle tenderness as the dependent variable and the following as the independent variables: Current migraine, Days until next migraine attack, days since last migraine attack, Sleep quality, physical activity, stiff neck (subjective feeling).
  The result shows how much of the variability in muscle hardness that can be explained by the independent variables.

SECONDARY OUTCOMES:
Day to day variation of muscle hardness in non-headache days | Daily measurements for about 30-60 days in a row
  Muscle hardness will be measured every day with Ultrasound elastography. Migraine and headache is noted in a headache diary.
Day to day variation of muscle tenderness in non-headache days | Daily measurements for about 30-60 days in a row
  Muscle tenderness will be measured every day with pressure pain threshold. Migraine and headache is noted in a headache diary.
Prodromes in migraine patients assessed by self-reported questionnaires | Patients are every day asked of symptoms for the last 24 hours and current symptoms
  Descriptive data of how often migraine patients experience prodrome like symptoms
Effect of tension type headache on muscle hardness | Daily measurements for about 30-60 days in a row
  Muscle hardness will be measured every day with Ultrasound elastography. Migraine and headache is noted in a headache diary.
  Is the measurements performed on headache days higher than those with out temporal proximity to headache.
Effect of tension type headache on muscle tenderness. | Daily measurements for about 30-60 days in a row
  Muscle tenderness will be measured every day with pressure pain threshold. Migraine and headache is noted in a headache diary.
  Is the measurements performed on headache days higher than those with out temporal proximity to headache.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided